CLINICAL TRIAL: NCT05536284
Title: Potential Drug Interactions With Bisoprolol in Egyptian Patients With Acute Coronary Syndrome
Brief Title: Potential Drug Interactions With Bisoprolol in Egyptian Patients With ACS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BisoprololDDI
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Acute coronary syndrome patients (Experimental): Acute coronary syndrome patients that are prescribes bisoprolol
  Interventions: Drug: Bisoprolol Fumarate Tablets

INTERVENTIONS:
Drug: Bisoprolol Fumarate Tablets — Antihypertensive drug used for acute coronary syndrome patients
  Other Names: concor

SUMMARY:
Acute coronary syndrome (ACS) is any group of clinical symptoms compatible with acute myocardial ischemia and includes unstable angina (UA), non-ST-segment elevation myocardial infarction (NSTEMI), and ST-segment elevation myocardial infarction (STEMI). (1). In Egypt, the overall prevalence of coronary heart disease (CHD) is 8.3 % (2). In addition, CHD in Egypt is the principal cause of death, responsible for 21.73% of total mortality (2).

Beta-blockers have shown to reduce the short-term risk of a reinfarction and the long-term risk of all-cause mortality and cardiovascular mortality (3). Beta blockers are used within 24 hours of ACS and given as long-term therapy after discharge (4). The Most frequently used drug in Egypt is bisoprolol. In patients with myocardial infarction undergoing primary percutaneous coronary intervention, early intravenous betablocker before reperfusion reduced infarct size and increased left ventricular ejection fraction (4).drug interactions are common in ACS patients due to polypharmacy and comorbidities.(5) there are limited studies investigating drug interactions with bisoprolol in acute coronary syndrome patients. The proposed research in this application will investigate potential drug interactions with bisoprolol in patients with acute coronary syndrome.

DETAILED DESCRIPTION:
1. Ethical committee approval will be obtained from Ethics committee of Faculty of Pharmacy, Damanhour University.
2. All participants should agree to take part in this clinical study and will provide informed consent.
3. Over 100 patients diagnosed with acute coronary syndrome for whom bisoprolol therapy is prescribed , will be recruited from Alexandria university hospital.
4. Blood samples for plasma concentration measurements of bisoprolol will be drawn at steady-state peak levels after 2-4 hours of administration of bisoprolol.

6. Heart rate and blood pressure of the patients will be measured to assess the clinical effect of bisoprolol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted with chest pain suspected to have ACS (acute coronary syndrome).
2. Both with ST elevation (STEMI) and without ST elevation (N-STEMI ) and unstable angina.
3. indicated to bisoprolol therapy

Exclusion Criteria:

Patients with contraindications to Bisoprolol therapy:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Bisoprolol peak level | 6 months
  Bisoprolol peak concentration level

CONTACTS AND LOCATIONS:
Overall Officials: Amira B Kassem, PHD, Study Director — Lecturer of Clinical Pharmacy, Damanhour University.; sherouk okda, bachelor, Principal Investigator — Clinical Pharmacy Specialist, Damanhour University.; Noha ahmed, PHD, Study Chair — Lecturer of Clinical Pharmacy, Damanhour University.; ahmad salahaldin, PHD, Study Director — Lecturer of biochemisrty, Damanhour University.; ahmad alamrawy, PHD, Study Chair — cardiologist , alexandria university; sohila alonsy, PHD, Study Chair — Lecturer of Analytical chemistry, Damanhour University.
Locations (1):
- Damanhour University, Damanhur, Beheira, Egypt

IPD SHARING:
Plan to Share IPD: No
The summary of all relevant data

REFERENCES:
- [Background] Almahmeed W, Arnaout MS, Chettaoui R, Ibrahim M, Kurdi MI, Taher MA, Mancia G. Coronary artery disease in Africa and the Middle East. Ther Clin Risk Manag. 2012;8:65-72. doi: 10.2147/TCRM.S26414. Epub 2012 Feb 16. PMID 22368447
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] Ibanez B, Macaya C, Sanchez-Brunete V, Pizarro G, Fernandez-Friera L, Mateos A, Fernandez-Ortiz A, Garcia-Ruiz JM, Garcia-Alvarez A, Iniguez A, Jimenez-Borreguero J, Lopez-Romero P, Fernandez-Jimenez R, Goicolea J, Ruiz-Mateos B, Bastante T, Arias M, Iglesias-Vazquez JA, Rodriguez MD, Escalera N, Acebal C, Cabrera JA, Valenciano J, Perez de Prado A, Fernandez-Campos MJ, Casado I, Garcia-Rubira JC, Garcia-Prieto J, Sanz-Rosa D, Cuellas C, Hernandez-Antolin R, Albarran A, Fernandez-Vazquez F, de la Torre-Hernandez JM, Pocock S, Sanz G, Fuster V. Effect of early metoprolol on infarct size in ST-segment-elevation myocardial infarction patients undergoing primary percutaneous coronary intervention: the Effect of Metoprolol in Cardioprotection During an Acute Myocardial Infarction (METOCARD-CNIC) trial. Circulation. 2013 Oct 1;128(14):1495-503. doi: 10.1161/CIRCULATIONAHA.113.003653. Epub 2013 Sep 3. PMID 24002794
- [Background] Taguchi M, Nozawa T, Igawa A, Inoue H, Takesono C, Tahara K, Hashimoto Y. Pharmacokinetic variability of routinely administered bisoprolol in middle-aged and elderly Japanese patients. Biol Pharm Bull. 2005 May;28(5):876-81. doi: 10.1248/bpb.28.876. PMID 15863897
- [Background] Tjandrawinata RR, Setiawati E, Yunaidi DA, Santoso ID, Setiawati A, Susanto LW. Bioequivalence study of two formulations of bisoprolol fumarate film-coated tablets in healthy subjects. Drug Des Devel Ther. 2012;6:311-6. doi: 10.2147/DDDT.S36567. Epub 2012 Oct 30. PMID 23139624
- [Background] Abolbashari M, Macaulay TE, Whayne TF, Mukherjee D, Saha S. Polypharmacy in Cardiovascular Medicine: Problems and Promises! Cardiovasc Hematol Agents Med Chem. 2017 Nov 8;15(1):31-39. doi: 10.2174/1871525715666170529093442. PMID 28552061